CLINICAL TRIAL: NCT06727903
Title: Development of a Predictive Model for Mortality in Patients Aged 75 or Older With Critical Illness
Brief Title: Predictive Model for Mortality in Older People With Critical Illness
Acronym: VITA
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-66
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness
Keywords: Critical Illness; Mortality; Aged; Intensive Care Units
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: laboratory biomarker analysis — Results of laboratory biomarker analysis will be analyzed as predictors for mortality

SUMMARY:
The present study aims to develop a predictive model to identify elderly patients with the highest likelihood of mortality upon admission to an intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 75 or older.
* Admission to an ICU from the Emergency Department.
* Availability of or possibility to contact a participant's informant.
* Informed consent for participation in the study, either by the participant or a valid legal representative.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria will not be included in the study:

* Patients transferred to the Emergency Department from a hospital ward.
* Patients who die within the first 24 hours of ICU admission.
* Patients admitted to Step-Down Units.
* Patients requiring ICU admission for any of the following reasons:

Orotracheal intubation or advanced cardiopulmonary resuscitation performed prior to arrival at the Emergency Department.

AV block awaiting pacemaker implantation. Activation of the STEMI or Stroke care pathway. Post-cardiac catheterization for acute coronary syndrome.

* Participation in another clinical study involving an intervention, procedure, or visit schedule that is incompatible with the present study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to a Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
mortality | Day 90
  mortality on day 90 from admission to Intensive Care Unit

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Hospital German Trias i Pujol, Badalona, Barcelona
  - Consorci Sanitari Alt Penedès-Garraf, Sant Pere de Ribes, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de Mataró, Barcelona
  - Hospital de Terrassa, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Dexeus Barcelona, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital General de Granollers, Barcelona
  - Hospital Sagrat Cor, Barcelona
  - Clinica Girona, Girona
  - Hospital Santa Caterina, Girona
  - Hospital Universitari Dr. Josep Trueta, Girona

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.